CLINICAL TRIAL: NCT03867461
Title: Prospective Measurement of Blood Pressure and End Tidal Carbon Dioxide Content Effects on Venous Sinus Caliber and Pressures in Patients With Idiopathic Intracranial Hypertension Undergoing Stenting
Brief Title: The Effects of MAP and EtCO2 on Venous Sinus Pressures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00055942
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-04

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: End-Tidal Carbon Dioxide; Venous Sinus Stenting; Venous Sinus Caliber and Pressures
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): Adult patients determined to be candidates for venous sinus stenting.
  End tidal CO and Mean Arterial Pressure will be adjusted to the following parameters during the intervention:
  For Group A: Initial Recording: Mean Arterial Pressure 60-80 mmHg, End tidal CO2 38-40 mmHg, Subsequent Recording: Mean Arterial Pressure 100-80 mmHg, End tidal CO2 38-40 mmHg.
  Interventions: Procedure: Venous Sinus Stenting; Other: Adjustment to end-tidal carbon dioxide concentrations ( 38-40 mmHg range); Other: Adjustment to Mean Arterial Pressure (100-110 mmHg range)
- Group B (Active Comparator): Adult patients determined to be candidates for venous sinus stenting.
  End tidal CO and Mean Arterial Pressure will be adjusted to the following parameters during the intervention:
  For Group B: Initial Recording: Mean Arterial Pressure 100-110 mmHg, End tidal CO2 38-40 mmHg, Subsequent Recording: Mean Arterial Pressure 60-80 mmHg, End tidal CO2 38-40 mmHg,
  Interventions: Procedure: Venous Sinus Stenting; Other: Adjustment to end-tidal carbon dioxide concentrations ( 38-40 mmHg range); Other: Adjustment to Mean Arterial Pressure (60-80 mmHg range)
- Group C (Active Comparator): Adult patients determined to be candidates for venous sinus stenting.
  End tidal CO and Mean Arterial Pressure will be adjusted to the following parameters during the intervention:
  For Group C: Initial Recording: Mean Arterial Pressure 100-110 mmHg, End tidal CO2 24-26 mmHg, Subsequent Recording: Mean Arterial Pressure 100-110 mmHg, End tidal CO2 38-40 mmHg,
  Interventions: Procedure: Venous Sinus Stenting; Other: Adjustment to end-tidal carbon dioxide concentrations ( 38-40 mmHg range); Other: Adjustment to Mean Arterial Pressure (100-110 mmHg range)
- Group D (Active Comparator): Adult patients determined to be candidates for venous sinus stenting.
  End tidal CO and Mean Arterial Pressure will be adjusted to the following parameters during the intervention:
  For Group D: Initial Recording: Mean Arterial Pressure 100-110 mmHg, End tidal CO2 38-40 mmHg, Subsequent Recording: Mean Arterial Pressure 100-100 mmHg, End tidal CO2 24-24 mmHg,
  Interventions: Procedure: Venous Sinus Stenting; Other: Adjustment to Mean Arterial Pressure (100-110 mmHg range); Other: Adjustment to end-tidal carbon dioxide concentrations (24-26 mmHg range)

INTERVENTIONS:
Procedure: Venous Sinus Stenting — Venous sinus stenting is performed under general anesthesia. Patients are loaded with aspirin and clopidogrel before the procedure. After induction, the right femoral vein is accessed and an 8 F sheath is placed. Intravenous heparin is administered. A 0.070-0.088 guide catheter is navigated into the ipsilateral jugular vein near the jugular bulb. Pre-stenting manometry is performed in every patient. To do so, a Renegade Hi-Flo microcatheter is navigated into the superior sagittal sinus and then used to measure ipsilateral venous pressures across the site of outflow obstruction (this will be the time point where the study intervention will be performed).
Other: Adjustment to end-tidal carbon dioxide concentrations ( 38-40 mmHg range) — End-tidal carbon dioxide concentrations will be adjusted to fall in the End-tidal carbon dioxide concentrations will be adjusted to fall in the 38-40 mmHg range
  Arms: Group A; Group B; Group C
Other: Adjustment to Mean Arterial Pressure (100-110 mmHg range) — Mean arterial pressure will be adjusted to fall in the 100-110 mmHg range
  Arms: Group A; Group C; Group D
Other: Adjustment to Mean Arterial Pressure (60-80 mmHg range) — Mean arterial pressure will be adjusted to fall in the 60-80 mmHg range
  Arms: Group B
Other: Adjustment to end-tidal carbon dioxide concentrations (24-26 mmHg range) — End-tidal carbon dioxide concentrations will be adjusted to fall in the 24-26 mmHg range
  Arms: Group D

SUMMARY:
The purpose of this study is to further elaborate the role of both arterial blood pressure and end-tidal carbon dioxide concentration on measured venous pressures.

DETAILED DESCRIPTION:
To prospectively evaluate the effect of changes in end-tidal carbon dioxide and arterial blood pressure on venous sinus pressure measurements in patients undergoing venous sinus stenting under general anesthesia. Venous sinus pressure measurements will increase with increases in both arterial blood pressure and end-tidal carbon dioxide concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Adults determined to be candidates for venous sinus stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Venous Sinus Pressures | Baseline
Venous Sinus Pressures | After intervention, up to 5 minutes

SECONDARY OUTCOMES:
Venous Sinus Diameter | Baseline
Venous Sinus Diameter | After Intervention, up to 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Fargen, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Satti SR, Leishangthem L, Chaudry MI. Meta-Analysis of CSF Diversion Procedures and Dural Venous Sinus Stenting in the Setting of Medically Refractory Idiopathic Intracranial Hypertension. AJNR Am J Neuroradiol. 2015 Oct;36(10):1899-904. doi: 10.3174/ajnr.A4377. Epub 2015 Aug 6. PMID 26251432
- [Background] Teleb MS, Cziep ME, Lazzaro MA, Gheith A, Asif K, Remler B, Zaidat OO. Idiopathic Intracranial Hypertension. A Systematic Analysis of Transverse Sinus Stenting. Interv Neurol. 2013;2(3):132-143. doi: 10.1159/000357503. PMID 24999351
- [Background] Levitt MR, Albuquerque FC, Gross BA, Moon K, Jadhav AP, Ducruet AF, Crowley RW. Venous sinus stenting in patients without idiopathic intracranial hypertension. J Neurointerv Surg. 2017 May;9(5):512-515. doi: 10.1136/neurintsurg-2016-012405. Epub 2016 May 19. PMID 27199383
- [Background] Ahmed RM, Wilkinson M, Parker GD, Thurtell MJ, Macdonald J, McCluskey PJ, Allan R, Dunne V, Hanlon M, Owler BK, Halmagyi GM. Transverse sinus stenting for idiopathic intracranial hypertension: a review of 52 patients and of model predictions. AJNR Am J Neuroradiol. 2011 Sep;32(8):1408-14. doi: 10.3174/ajnr.A2575. Epub 2011 Jul 28. PMID 21799038
- [Background] West JL, Garner RM, Greeneway GP, Traunero JR, Aschenbrenner CA, Singh J, Wolfe SQ, Fargen KM. Venous waveform morphological changes associated with treatment of symptomatic venous sinus stenosis. J Neurointerv Surg. 2018 Nov;10(11):1108-1113. doi: 10.1136/neurintsurg-2018-013858. Epub 2018 Mar 21. PMID 29563210
- [Background] Fargen KM, Spiotta AM, Hyer M, Lena J, Turner RD, Turk AS, Chaudry I. Comparison of venous sinus manometry gradients obtained while awake and under general anesthesia before venous sinus stenting. J Neurointerv Surg. 2017 Oct;9(10):990-993. doi: 10.1136/neurintsurg-2016-012608. Epub 2016 Sep 15. PMID 27634954
- [Background] Raper DMS, Buell TJ, Chen CJ, Ding D, Starke RM, Liu KC. Intracranial venous pressures under conscious sedation and general anesthesia. J Neurointerv Surg. 2017 Oct;9(10):986-989. doi: 10.1136/neurintsurg-2017-012984. Epub 2017 Mar 30. PMID 28360352
- [Background] West JL, Garner RM, Traunero JR, Wolfe SQ, Fargen KM. Changes in End-Tidal Carbon Dioxide Partial Pressure Alter Venous Sinus Pressure Measurements in Idiopathic Intracranial Hypertension. World Neurosurg. 2018 Dec;120:495-499. doi: 10.1016/j.wneu.2018.09.117. Epub 2018 Sep 26. PMID 30266712

DOCUMENTS (1):
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03867461/ICF_000.pdf